CLINICAL TRIAL: NCT02443675
Title: Observational Study of Pain Reduction in Late-Stage Cancer Patients Who Are Receiving Low-Dose Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cure Cancer Worldwide, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: C4 OS-1
Record Dates: First submitted 2015-05-02; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational Study of Pain Reduction in Late Stage Cancer Patients Receiving Low-Dose Chemotherapy

DETAILED DESCRIPTION:
Observational Study of Pain Reduction in Late Stage Cancer Patients who are Receiving Low-Dose Chemotherapy (Metabolic Targeting)

ELIGIBILITY:
Inclusion Criteria:

* Patient requests to be included in this study

Exclusion Criteria:

* Patient does not request to be included in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients Receiving Low Dose Chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pain Level Self Assessment | 5 years
  From enrollment in study to termination of study (August 2020)

CONTACTS AND LOCATIONS:
Overall Officials: gary l smith, mba, Study Director — Cure Cancer Worldwide, LLC